CLINICAL TRIAL: NCT04401020
Title: An Open-label, First-in-human, Single Agent, Dose Escalation Study for the Evaluation of Safety, Pharmacokinetics, Pharmacodynamics and Anti-tumor Activity of SAR442257 in Patients With Relapsed and Refractory Multiple Myeloma and Relapsed and Refractory Non-Hodgkin Lymphoma
Brief Title: First-in-human Single Agent Study of SAR442257 in RRMM and RR-NHL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TED16364; U1111-1244-2511 (Registry Identifier: UTN); 2023-508358-24 (Registry Identifier: CTIS); 2019-003390-26 (EudraCT Number)
Record Dates: First submitted 2020-05-12; First posted 2020-05-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation (Experimental): SAR442257 will be given intravenously with lead-in doses (LID) in the first-week, followed by once weekly until week 4 (Cycle 1) and once weekly for each subsequent cycle(s).
  Interventions: Drug: SAR442257

INTERVENTIONS:
Drug: SAR442257 — Pharmaceutical form: Sterile powder for reconstitution Route of administration: Intravenous infusion

SUMMARY:
Primary Objective:

To determine the maximum tolerated dose (MTD) of SAR442257 administered as a single agent in patients with relapsed and refractory multiple myeloma (RRMM) and relapsed and refractory non-Hodgkin lymphoma (RR-NHL), and determine the recommended Phase 2 dose (RP2D)

Secondary Objectives:

* To characterize the safety profile of SAR442257
* To characterize the pharmacokinetics (PK) profile of SAR442257
* To assess preliminary evidence of antitumor activity

DETAILED DESCRIPTION:
Study duration per participant is 2 months to estimated 16 months. Cycle lengths in this study are 27 days in Cycle 1 and 28 days for subsequent cycles as determined by totality of data collected thus far including PK/Pharmacodynamics (PD), safety and preliminary efficacy.

ELIGIBILITY:
Inclusion criteria :

Participant must be at least 18 years of age or of the country's legal age of majority if the legal age is >18 years old, at the time of signing the informed consent.

Life expectancy of at least 12 weeks. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.

RRMM patients:

must have received at least 3 prior lines of therapy including proteasome inhibitor (PI), immunomodulatory agent (IMiD), and anti-CD38 mAb;

and must be refractory to anti-CD38 antibody (eg, daratumumab or isatuximab), characterized by progression within 60 days of the last dose of anti-CD38, regardless of which line it was given; and must be either relapsed or refractory to all established therapies with known clinical benefit in RRMM where approved and available, or are intolerant to those established therapies; based upon investigator's clinical judgement.

and must not be candidates for regimens known to provide clinical benefit based upon investigator's clinical judgement.

Patients with RRMM must have measurable disease as per the following:

* Serum M protein ≥0.5 g/dL (≥5 g/L), or
* Urine M protein ≥200 mg/24 hours, or
* Serum free light chain (FLC) assay: involved FLC assay ≥10 mg/dL and an abnormal serum FLC ratio (<0.26 or >1.65).

Patients with RR-NHL must be relapsed or refractory to all established therapies with known clinical benefit where approved and available, or are intolerant to those established therapies; based upon investigator's clinical judgement.

Patients with RR-NHL must have measurable disease of at least one lesion ≥1.5 cm as documented by computed tomography (CT) scan, including the following subtype of disease:

* Diffuse large B-cell lymphoma (DLBCL).
* HGBCL with MYC and/or BCL2 and/or BCL6 rearrangement or HGBCL NOS,
* transformed follicular lymphoma (tFL),
* follicular lymphoma (FL),
* mantle cell lymphoma (MCL),
* marginal zone lymphoma (MZL),
* lymphoplasmacytic lymphoma,
* small lymphocytic lymphoma (SLL). Patients with RR-NHL subtype T cell lymphoma (TCL) including the following subtype of disease: Nodal peripheral TCL including angio-immunoblastic TCL (AITL), anaplastic large cell lymphoma (ALCL), adult T cell leukemia-lymphoma, and peripheral TCL NOS (not otherwise specified). Peripheral TCL of the innate immune system: breast implant ALCL, extranodal NK/TCL, enteropathy associated TCL, monomorphic epitheliotropic intestinal TCL, and hepatosplenic TCL. histopathologically confirmed mycosis fungoides or Sézary syndrome (cutaneous T cell lymphoma [CTCL] stage IIB or greater according to the European Organization for Research and Treatment of Cancer/International Society for Cutaneous Lymphomas [EORTC-ISCL] consensus classification) at study entry with progressive, persistent, or recurrent disease who have no available remaining standard therapeutic options (ie, refractory) as determined by the Investigator.

Patients with lymphoma must have availability of lymphoma tissue for biomarker testing: either archived tissue or a fresh biopsy as a part of screening. On-treatment biopsy (Cycle 2 or beyond) is also expected if disease location is in a superficial lymph node. For post-CAR-T patients a fresh LN biopsy is expected if in a superficial node. For these patients tissue materials should be made available for analysis during the study. Excisional biopsy or resected tissue is required if clinically feasible; otherwise, core needle biopsy is acceptable. Fine needle aspirates are not acceptable.

Patients with lymphoma must have a ≥50% left ventricular ejection fraction (LVEF) and no pericardial effusion, as measured by echocardiogram (ECHO).

Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion criteria:

Diagnosed or treated for another malignancy within 3 years prior to enrollment, except for basal cell carcinoma or squamous cell carcinoma of the skin, an in-situ malignancy, superficial bladder carcinoma or low risk prostate cancer.

Amyloidosis, chronic lymphocytic leukemia and prolymphocytic leukemia. Known central nervous system (CNS) involvement by myeloma, lymphoma or other CNS disease such as neurodegenerative condition or CNS movement disorder.

Has congestive heart failure (New York Heart Association) Grade ≥II; cardiomyopathy, active ischemia, or any other uncontrolled cardiac condition such as angina pectoris, clinically significant arrhythmia requiring therapy including anticoagulants, or clinically significant uncontrolled hypertension, QT interval corrected by the Fridericia method >480 msec (Grade ≥2). Acute myocardial infarction within 6 months before start of study treatment.

Has active autoimmune disease including autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura, inflammatory bowel syndrome, pneumonitis or any chronic condition requiring a higher corticosteroid systemic equivalent than prednisone 10 mg daily.

Clinically-not controlled chronic or ongoing infectious disease requiring treatment at the time of first dose or within the 14 days before first dose.

Active hepatitis A, B, and C as defined below: active hepatitis A (defined as positive IgM), active hepatitis B (defined as either positive hepatitis B surface antigen or positive hepatitis B viral DNA test above the lower limit of detection of the assay, and hepatitis B core antibodies), or C infection (defined as a known positive hepatitis C antibody result and known quantitative hepatitis C [HCV] ribonucleic acid [RNA] results greater than the lower limits of detection of the assay).

Known positivity for Human Immunodeficiency Virus (HIV). Unresolved toxicities from prior anticancer therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade 1 or to levels dictated in the eligibility criteria with the exception of Grade 1 peripheral neuropathy, alopecia or toxicities from prior anticancer therapy that are considered irreversible (defined as having been present and stable for >4 weeks) which may be allowed if they are not otherwise described in the exclusion criteria.

Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD) | Baseline to estimated 4 weeks
  MTD: defined as the highest dose level (DL) with highest probability of Investigational Medicinal Product (IMP)-related dose limiting toxicity (DLT) rate within the target range (16 to 33%) among dose levels with less than 0.25 probability of DLT rate above target (>33%)
Determine recommended Phase 2 dose (RP2D) | Baseline to estimated 4 months
  RP2D: defined as the dose selected for the further single agent testing in the future study

SECONDARY OUTCOMES:
Number of participants with AEs/SAEs/AESI | Baseline to 30 days after end of treatment
  Incidence of treatment-emergent adverse events (AEs)/serious adverse events (SAEs)/ adverse events of special interest (AESIs) and laboratory abnormalities
Assessment of pharmacokinetic (PK) parameter: Cmax | through study completion (estimated 16 months)
  Maximum concentration observed (Cmax)
Assessment of PK parameter: Ctrough | through study completion (estimated 16 months)
  Concentration observed just before treatment administration during repeated dosing (Ctrough)
Assessment of PK parameter: AUC0-τ | up to 4 weeks
  Area under the concentration versus time curve during a dosing interval (T) (AUC0-τ)
Overall response rate for RRMM | Baseline to 6 months
  Overall response rate will be assessed using the International Myeloma Working Group (IMWG) 2016 criteria for patients with RRMM
Overall response rate for RR-NHL | Baseline to 6 months
  Overall response rate will be assessed using the Response evaluation criteria in lymphoma (RECIL) 2017 criteria for patients with RR-NHL

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- United States (3):
  - City of Hope Site Number : 8400001, Duarte, California
  - University of Miami - Sylvester Comprehensive Cancer Center Site Number : 8400005, Miami, Florida
  - Mayo Clinic of Rochester Site Number : 8400003, Rochester, Minnesota
- Czechia (3):
  - Investigational Site Number : 2030003, Brno
  - Investigational Site Number : 2030001, Ostrava - Poruba
  - Investigational Site Number : 2030002, Prague
- Norway (2):
  - Investigational Site Number : 5780001, Oslo
  - Investigational Site Number : 5780101, Oslo
- South Korea (2):
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (6):
  - Investigational Site Number : 7240005, Santander, Cantabria
  - Investigational Site Number : 7240003, Badalona, Catalunya [Cataluña]
  - Investigational Site Number : 7240006, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240001, Pamplona, Navarre
  - Investigational Site Number : 7240007, Madrid
  - Investigational Site Number : 7240004, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org